CLINICAL TRIAL: NCT04310371
Title: Exposure to CARDIovascular Risk Assessed by Cardiac Adiposity in oBese adOlescents Eligible to a Residential Long-term Lifestyle Intervention by Diet and eXercise
Brief Title: Exposure to CARDIovascular Risk Assessed by Cardiac Adiposity in oBese adOlescents Eligible to a Residential Long-term Lifestyle Intervention by Diet and eXercise (CARDIBOX)
Acronym: CARDIBOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other); LaPSCo laboratory, Physiological and Psychosocial Stress, UMR CNRS 6024, Clermont-Ferrand, France (Unknown); LaPEC laboratory (EA 4278), University of Avignon, Avignon, France (Unknown); Child Medical Center, 3 Rue de la Prugne, 63540 Romagnat, France (Unknown); Tza-Nou Center, 230 Rue Vercingétorix, 63150 La Bourboule, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2019 DUTHEIL; 2019-A01804-53 (Other: ANSM)
Record Dates: First submitted 2020-02-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Adolescent Obesity
Keywords: left myocardial regional function; cardiac ectopic fat deposits; lifestyle programm; prevention; Adolescent Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: participants receive an intervention throughout the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese adolescents (Experimental): BMI greater than the 97th percentile of national curves. Participants will follow a 3-month lifestyle intervention
  Interventions: Behavioral: 3-month lifestyle intervention
- Control group (No Intervention): to be normal-weighted (no obesity if overweight, <85th percentile of national curves).

INTERVENTIONS:
Behavioral: 3-month lifestyle intervention — Adolescents from the intervention group will be enrolled at the obesity center for the whole school year (i.e., 10 months). The physical activity program consists of two training sessions (aerobic and resistance training) per week.
  There will be two measurement time: one at baseline (Day 0) and one at three months after the beginning of the lifestyle intervention (M3). The controls will be evaluated at baseline only.
  Arms: Obese adolescents

SUMMARY:
The high prevalence of childhood obesity is a major public health issue, worldwide. Childhood obesity is associated with a high risk of cardiovascular events in adulthood, but recent studies also point out the development of cardiovascular complications in childhood or adolescence justifying the need for early detection and appropriate therapeutic management to prevent the development of more severe abnormalities. This project proposes to evaluate the myocardial function in a fine and comprehensive way (longitudinal, circumferential and radial linear deformations, and rotation / torsion mechanics) from the deformation imaging (MRI and high-resolution echocardiography), in obese adolescents following a lifestyle intervention combining diet and physical activity.

DETAILED DESCRIPTION:
The investigators aim to improve knowledge of the association between epicardial adipose tissue, myocardial lipid content, and left ventricular regional myocardial function.

In this protocol, obese adolescents are recruited undergoing a 3-month lifestyle intervention residential program. Adolescents from the intervention group will be enrolled at the obesity center for the whole school year. The obesity center employs a multidisciplinary team to provide the best weight management care to adolescents during their stay. The weight loss program is an integral part of the obesity center program and fundamentally combines physical activity with a normocaloric diet monitored by a dietician. The physical activity program consists of two training sessions (aerobic and resistance training) per week. Moreover, adolescents will be engaged in two additional sessions per week, consisting in recreational activities such as ball and racquet games, trekking, snowshoeing or swimming.

There will be two measurement time: one at baseline (Day 0) and one at three months after the beginning of the lifestyle intervention (M3). The controls will be evaluated at baseline only.

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be two-sided and p inferior to 0.05 will be considered significant. Qualitative variables will be described in terms of numbers and proportions. Quantitative variables will be described in terms of numbers, mean standard deviation or median according to statistical distribution (normality studied using Shapiro-Wilk test). Graphic representations will be complete presentations of results. The main analysis will be performed with the Stata software (version 13, StataCorp, College Station). All statistical tests will be carried out at a risk of error of first species α set at 5%. Most of the analysis of the secondary evaluation criteria will be exploratory in nature and may lack power in terms of numbers. As discussed by Feise in 2002,104 the adjustment of the risk of error of 1st species will not be systematically proposed, but case by case in view of clinical considerations and not only statistical (e.g. Sidak correction for the analysis of correlation coefficients).

Qualitative variables will be described in terms of numbers and proportions. Quantitative variables will be described in terms of standard deviation or mean median according to statistical distribution (normality studied using Shapiro-Wilk test). Graphic representations will be complete presentations of results.

Intergroup comparisons will be systematically conducted without adjustment and by adjusting for factors whose distribution could be unbalanced between groups. Patients will be described and compared between groups at inclusion according to the following variables: compliance with eligibility criteria, epidemiological characteristics, clinical characteristics and characteristics of possible treatments. The baseline comparability of the two groups will be assessed on the main characteristics of the participants and potential factors associated with the primary outcome. A possible difference between the two groups on one of these characteristics will be determined according to clinical considerations and not solely statistical ones.

ELIGIBILITY:
Inclusion Criteria:

* age between 12 and 16 years old
* mature (menarche)
* suitable for physical activity
* able to give an informative consent
* affiliated at French insurance company
* consent from the legal representatives
* For obese adolescents: BMI greater than the 97th percentile of national curves.
* For the control group: to be normal-weighted (no obesity if overweight, <85th percentile of national curves).

Exclusion Criteria:

* Medical or surgical history judged by the investigator as incompatible with the study
* Drugs that may interfere with the study results
* Cardiovascular, hepatic, psychiatric, renal, or endocrinological diseases
* Smoking
* Alcohol consumption
* Intense physical activity in competition

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
cardiac ectopic fat deposits | Month 3
  Quantification of cardiac ectopic fat deposits (thickness using echocardiography)
cardiac ectopic fat deposits | Day 0
  Quantification of cardiac ectopic fat deposits (thickness using echocardiography)
cardiac ectopic fat deposits | Day 0
  Quantification of cardiac ectopic fat deposits (volume using MRI)
cardiac ectopic fat deposits | Month 3
  Quantification of cardiac ectopic fat deposits (volume using MRI)
cardiac ectopic fat deposits | Month 3
  Quantification of cardiac ectopic fat deposits (myocardial triglyceride content evaluated by MRI)
cardiac ectopic fat deposits | Day 0
  Quantification of cardiac ectopic fat deposits (myocardial triglyceride content evaluated by MRI)
left myocardial regional function | Month 3
  left myocardial regional function (echocardiography)
left myocardial regional function | Month 3
  left myocardial regional function (MRI)
left myocardial regional function | Day 0
  left myocardial regional function (echocardiography)
left myocardial regional function | Day 0
  left myocardial regional function (MRI)

SECONDARY OUTCOMES:
macrovascularisation | Day 0
  measure of carotid intima-media thickness (CIMT) using High-resolution B-mode ultrasound
macrovascularisation | Month 3
  measure of carotid intima-media thickness (CIMT) using High-resolution B-mode ultrasound
microvascularisation | Month 3
  measure of blood flow velocity using laser speckle contrast imaging (LSCI)
microvascularisation | Day 0
  measure of blood flow velocity using laser speckle contrast imaging (LSCI)
microvascularisation | Day 0
  measure of microvascular perfusion using laser-Doppler flowmetry (LDF)
microvascularisation | Month 3
  measure of microvascular perfusion using laser-Doppler flowmetry (LDF)
microvascularisation | Month 3
  measure of microvascular perfusion using Iontophoresis procedure
microvascularisation | Day 0
  measure of microvascular perfusion using Iontophoresis procedure
microvascularisation | Day 0
  measure of microvascular perfusion using flowmotion
microvascularisation | Month 3
  measure of microvascular perfusion using flowmotion
heart rate variability | Month 3
  measure of heart rate variability using a holter
heart rate variability | Day 0
  measure of heart rate variability using a holter
skin conductance | Day 0
  measure of skin conductance using Wristband electrodes - Empatica E4
skin conductance | Month 3
  measure of skin conductance using Wristband electrodes - Empatica E4
Liver steatosis | Month 3
  measure of liver steatosis by MRI
Liver steatosis | Day 0
  measure of liver steatosis by MRI
Liver steatosis | Day 0
  measure of liver steatosis by fibroscanner (ultrasonic attenuation)
Liver steatosis | Month 3
  measure of liver steatosis by fibroscanner (ultrasonic attenuation)
Liver steatosis | month 3
  measure of liver steatosis by Aixplorer (Lipersonic Imagine®)
Liver steatosis | Day 0
  measure of liver steatosis by Aixplorer (Lipersonic Imagine®)
Liver fibrosis | Day 0
  measure of liver fibrosis by fibroscanner (liver stiffness)
Liver fibrosis | Month 3
  measure of liver fibrosis by fibroscanner (liver stiffness)
Liver fibrosis | Month 3
  measure of liver fibrosis by fibrotest (Lipersonic Imagine®)
Liver fibrosis | Day 0
  measure of liver fibrosis by fibrotest (Lipersonic Imagine®)
blood pressure | Day0
  measure of blood pressure using sphygmomanometer
blood pressure | month 3
  measure of blood pressure using sphygmomanometer
Fitness | Month 3
  6-minutes walking test to assess functional capacity at a sub-maximal level, and the effects of exercise training in cardiac and pulmonary patients.
Fitness | Day 0
  6-minutes walking test to assess functional capacity at a sub-maximal level, and the effects of exercise training in cardiac and pulmonary patients.
muscle mass | Month 3
  measure of muscle mass using impedancemeter
fat mass | Month 3
  measure of muscle mass using impedancemeter
bone structure | Month 3
  measure of muscle mass using impedancemeter
muscle mass | Day 0
  measure of muscle mass using impedancemeter
fat mass | Day 0
  measure of muscle mass using impedancemeter
bone structure | Day 0
  measure of muscle mass using impedancemeter
muscle mass | Day 0
  measure of muscle mass using Densitometry X-ray absorption
fat mass | Day 0
  measure of muscle mass using Densitometry X-ray absorption
bone structure | Day 0
  measure of muscle mass using Densitometry X-ray absorption
muscle mass | Month 3
  measure of muscle mass using Densitometry X-ray absorption
fat mass | Month 3
  measure of muscle mass using Densitometry X-ray absorption
bone structure | Month 3
  measure of muscle mass using Densitometry X-ray absorption
muscle mass | Month 3
  measure of muscle mass using Peripheral quantitative computed tomography (pQCT)
fat mass | Month 3
  measure of muscle mass using Peripheral quantitative computed tomography (pQCT)
bone structure | Month 3
  measure of muscle mass using Peripheral quantitative computed tomography (pQCT)
muscle mass | Day 0
  measure of muscle mass using Peripheral quantitative computed tomography (pQCT)
fat mass | Day 0
  measure of muscle mass using Peripheral quantitative computed tomography (pQCT)
bone structure | Day 0
  measure of muscle mass using Peripheral quantitative computed tomography (pQCT)
muscle mass | Day 0
  measure of muscle mass using Quantitative ultrasounds (QUS)
fat mass | Day 0
  measure of muscle mass using Quantitative ultrasounds (QUS)
bone structure | Day 0
  measure of muscle mass using Quantitative ultrasounds (QUS)
muscle mass | Month 3
  measure of muscle mass using Quantitative ultrasounds (QUS)
fat mass | Month 3
  measure of muscle mass using Quantitative ultrasounds (QUS)
bone structure | Month 3
  measure of muscle mass using Quantitative ultrasounds (QUS)
depression | Day 0
  depression is assessed by the Hospital Anxiety and Depression scale (HAD) composed by 7 items and a 4-point scale from "never" to "always".
depression | Month 3
  depression is assessed by the Hospital Anxiety and Depression scale (HAD) composed by 7 items and a 4-point scale from "never" to "always".
anxiety | Day 0
  anxiety is assessed by the Hospital Anxiety and Depression scale (HAD) composed by 7 items and a 4-point scale from "never" to "always". It is also evaluated by the State-Trait Anxiety Inventory (STAI) composed by two dimensions, state anxiety and trait anxiety, both evaluated with a 20-items questionnaire on a 4-point scale from "never" to "always"
anxiety | Month 3
  anxiety is assessed by the Hospital Anxiety and Depression scale (HAD) composed by 7 items and a 4-point scale from "never" to "always". It is also evaluated by the State-Trait Anxiety Inventory (STAI) composed by two dimensions, state anxiety and trait anxiety, both evaluated with a 20-items questionnaire on a 4-point scale from "never" to "always"
General health | Day 0
  general health is assessed by the short form 36 health survey (SF36) composed by 36 items
General health | Month 3
  general health is assessed by the short form 36 health survey (SF36) composed by 36 items
Stress | day 0
  stress is assessed by a Visuel analog scale of 100mm ranging from very low (0) to very high (100)
Stress | Month 3
  stress is assessed by a Visuel analog scale of 100mm ranging from very low (0) to very high (100)
Fatigue | Day 0
  Fatigue is assessed by a Visuel analog scale of 100mm ranging from very low (0) to very high (100)
Fatigue | Month 3
  Fatigue is assessed by a Visuel analog scale of 100mm ranging from very low (0) to very high (100)
Sleep | day 0
  Burnout is assessed by the Maslach Burn-out Inventory (MBI) composed by 22 items and a 7-point scale ranging from "never" to "every day".
Sleep | Month 3
  Burnout is assessed by the Maslach Burn-out Inventory (MBI) composed by 22 items and a 7-point scale ranging from "never" to "every day".
Burnout | day 0
  Burnout is assessed by the Maslach Burn-out Inventory (MBI) composed by 22 items and a 7-point scale ranging from "never" to "every day".
Burnout | Month 3
  Burnout is assessed by the Maslach Burn-out Inventory (MBI) composed by 22 items and a 7-point scale ranging from "never" to "every day".
Mindfulness | Day 0
  Midfuless is assessed by the Freiburg Mindfulness Inventory-14 (FMI) composed by a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree)
Mindfulness | Month 3
  Midfuless is assessed by the Freiburg Mindfulness Inventory-14 (FMI) composed by a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree)
Coping | Day 0
  Coping is assessed by the Brief Illness Perception Questionnaire (B-IPQ) composed by an 11-point scale
Coping | Month 3
  Coping is assessed by the Brief Illness Perception Questionnaire (B-IPQ) composed by an 11-point scale
Emotions | Day 0
  Emotions are assessed by the Emotion Régulation Questionnaire (ERQ) composed by 10 items on a 7-point likert scale ranging from 1 (strongly disagree) to 7 (strongly agree)
Emotions | Month 3
  Emotions are assessed by the Emotion Régulation Questionnaire (ERQ) composed by 10 items on a 7-point likert scale ranging from 1 (strongly disagree) to 7 (strongly agree)
Perception of work | Day 0
  Work perception is assessed by the Job Demand-Control-Support (JDSC) questionnaire of Karasek composed by 26 items on a 4-point scale ranging from 1 (strongly disagree) to 4 (strongly agree). It is also evaluated by the effort-reward imbalance model (ERI) of Siegrist composed by 46 items on a 5-point scale ranging from 1 (no agreement) to 5 (agree and very disturb).
Perception of work | Month 3
  Work perception is assessed by the Job Demand-Control-Support (JDSC) questionnaire of Karasek composed by 26 items on a 4-point scale ranging from 1 (strongly disagree) to 4 (strongly agree). It is also evaluated by the effort-reward imbalance model (ERI) of Siegrist composed by 46 items on a 5-point scale ranging from 1 (no agreement) to 5 (agree and very disturb).
Self-efficacy | Day 0
  Self-efficacy is assessed by the perceived self-efficacy scale composed by 10 items on a 4-point scale
Self-efficacy | Month 3
  Self-efficacy is assessed by the perceived self-efficacy scale composed by 10 items on a 4-point scale
Alexithymia | Day 0
  Alexithymia is assessed by the Twenty-item Toronto Alexithymia Scale (TAS20) composed by a 5-point scale from "strongly agree" to "strongly disagree".
Alexithymia | Month 3
  Alexithymia is assessed by the Twenty-item Toronto Alexithymia Scale (TAS20) composed by a 5-point scale from "strongly agree" to "strongly disagree".
Illness perception | Day 0
  Perception of illness is assessed by the Brief Illness Perception Questionnaire (B-IPQ) composed by a 11-point scale.
Illness perception | Month 3
  Perception of illness is assessed by the Brief Illness Perception Questionnaire (B-IPQ) composed by a 11-point scale.
Metacognition | Day 0
  Metacognition is assessed by the MetaCognition Questionnaire (MCQ-30) composed by 30 items on a 5-point scale
Metacognition | Month 3
  Metacognition is assessed by the MetaCognition Questionnaire (MCQ-30) composed by 30 items on a 5-point scale
Time perception | Day 0
  Perception of the time is assessed by the Metacognitive questionnaire on time perception (MQT) composed by 24 items on a 5-point scale. It is also evaluated by the Zimbardo Time Perspective Inventory (ZPTI) composed by 56 items on a 5-point scale from "very uncharacteristic" to "very characteristic".
Time perception | Month 3
  Perception of the time is assessed by the Metacognitive questionnaire on time perception (MQT) composed by 24 items on a 5-point scale. It is also evaluated by the Zimbardo Time Perspective Inventory (ZPTI) composed by 56 items on a 5-point scale from "very uncharacteristic" to "very characteristic".
Physical activity | Day 0
  Physical activity is assessed by the Recent Physical Activity Questionnaire (RPAQ)
Physical activity | Month 3
  Physical activity is assessed by the Recent Physical Activity Questionnaire (RPAQ)
Life style | Day 0
  life style is assessed with a questionnaire on coffee consumption, food intake, etc
Life style | Month 3
  life style is assessed with a questionnaire on coffee consumption, food intake, etc
cholesterol | Day 0
  measure by blood analyses to evaluate alloplastic load
triglycerides | Day 0
  measure by blood analyses to evaluate alloplastic load
cholesterol | Month 3
  measure by blood analyses to evaluate alloplastic load
triglycerides | Month 3
  measure by blood analyses to evaluate alloplastic load
Cortisol | Day 0
  hormone measure by blood analyses to evaluate alloplastic load
Cortisol | Month 3
  hormone measure by blood analyses to evaluate alloplastic load
DHEAS | day 0
  hormone measure by blood analyses to evaluate alloplastic load
DHEAS | Month 3
  hormone measure by blood analyses to evaluate alloplastic load
BDNF | Day 0
  proteins measure by blood analyses to evaluate alloplastic load
BDNF | Month 3
  proteins measure by blood analyses to evaluate alloplastic load
CRP | Day 0
  proteins measure by blood analyses to evaluate alloplastic load
pro-inflammatory cytokines | Day 0
  proteins measure by blood analyses to evaluate alloplastic load
TNF alpha | Day 0
  proteins measure by blood analyses to evaluate alloplastic load
CRP | Month 3
  proteins measure by blood analyses to evaluate alloplastic load
pro-inflammatory cytokines | Month 3
  proteins measure by blood analyses to evaluate alloplastic load
TNF alpha | Month 3
  proteins measure by blood analyses to evaluate alloplastic load
NPY | Month 3
  proteins measure by blood analyses to evaluate alloplastic load
NPY | Day 0
  proteins measure by blood analyses to evaluate alloplastic load
Leptin | Day 0
  measure by blood analyses to evaluate appetite regulation
Leptin | Month 3
  measure by blood analyses to evaluate appetite regulation
Ghrelin | Day 0
  measure by blood analyses to evaluate appetite regulation
Ghrelin | Month 3
  measure by blood analyses to evaluate appetite regulation
NPY | day 0
  measure by blood analyses to evaluate appetite regulation
NPY | Month 3
  measure by blood analyses to evaluate appetite regulation
adiponectine | Day 0
  measure by blood analyses to evaluate appetite regulation
adiponectine | Month 3
  measure by blood analyses to evaluate appetite regulation
CCK | Day 0
  measure by blood analyses to evaluate appetite regulation
Month 3 | Day 0
  measure by blood analyses to evaluate appetite regulation
Insulin | Day 0
  measure by blood analyses to evaluate glucid metabolism
Insulin | Month 3
  measure by blood analyses to evaluate glucid metabolism
HbA1c | Day 0
  measure by blood analyses to evaluate glucid metabolism
HbA1c | Month 3
  measure by blood analyses to evaluate glucid metabolism
glucose | Day 0
  measure by blood analyses to evaluate glucid metabolism
glucose | Month 3
  measure by blood analyses to evaluate glucid metabolism
Albumin | Day 0
  measure by blood analyses to evaluate protid metabolism
Albumin | Month 3
  measure by blood analyses to evaluate protid metabolism
transthyretin | Day 0
  measure by blood analyses to evaluate protid metabolism
transthyretin | Month 3
  measure by blood analyses to evaluate protid metabolism
Homeostasis | Day 0
  measure of Fibroblast growth factor 23 (FGF23) by blood analyses to evaluate bone metabolism
Homeostasis | Month 3
  measure of Fibroblast growth factor 23 (FGF23) by blood analyses to evaluate bone metabolism
Osteoresorption | Day 0
  measure of C-terminal Telopeptide of Type I collagen (CTx) by blood analyses to evaluate bone metabolism
Osteoresorption | Month 3
  measure of C-terminal Telopeptide of Type I collagen (CTx) by blood analyses to evaluate bone metabolism
Osteoformation | Day 0
  measure of decarboxylated osteocalcine and BSAP by blood analyses to evaluate bone metabolism
Osteoformation | Month 3
  measure of decarboxylated osteocalcine and BSAP by blood analyses to evaluate bone metabolism
VEGF | Day 0
  measure by blood analyses to evaluate cardiovascular function
VEGF | Month 3
  measure by blood analyses to evaluate cardiovascular function
PAI1 | Day 0
  measure by blood analyses to evaluate cardiovascular function
PAI1 | Month 3
  measure by blood analyses to evaluate cardiovascular function
weight | Day 0
  measure of weight in kilograms
weight | Month 3
  measure of weight in kilograms
waist circumference | Day 0
  measure of waist circumference in centimetres
waist circumference | Month 3
  measure of waist circumference in centimetres

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided